CLINICAL TRIAL: NCT05540743
Title: The Efficacy of Anti-TNF Alpha Agents in the Treatment of JIA- Associated Uveitis in a Pediatric Cohort
Brief Title: Biologic Therapy in Pediatric JIA Uveitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mai Nasser Abd Elmohsen, lecturer of ophthalmology, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-50-2020
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Juvenile Idiopathic Arthritis Associated Uveitis
Keywords: Biologics; JIA-U; Uveitis; Pediatrics; adalimumab
MeSH Terms: conditions — Uveitis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- JIA associated uveitis (Other): patients diagnosed with Juvenile idiopathic arthritis and uveitis taking immunosuppression including biologics 9of any type according to their rheumatologist recommendations) for control of their autoimmune uveitis.
  Interventions: Drug: biologic DMARDs

INTERVENTIONS:
Drug: biologic DMARDs — follow up the clinical response in Egyptian population to the drug
  Other Names: rimicade, adalimumab

SUMMARY:
Juvenile Idiopathic Arthritis (JIA) remains the most common systemic disorder associated with pediatric uveitis. Studies estimate that 28-67% of patients with JIA-associated uveitis develop ocular complications, with 12% developing poor visual outcome. The only means of improving long term effects of uveitis, is early and aggressive anti-inflammatory treatment, including biologics.

DETAILED DESCRIPTION:
Juvenile Idiopathic Arthritis (JIA) remains, globally, the most common systemic disorder associated with pediatric uveitis consisting 75% of anterior uveitis cases (AU)1. In a cohort study from Cairo University Pediatric Hospital, JIA accounted for 39% of all cases of pediatric uveitis (unpublished data). Studies estimate that 28-67% of patients with JIA-U develop ocular complications, with 12% developing poor visual outcome2,3,4. Thus, early and aggressive anti-inflammatory treatment is the only means of improving long term effects of uveitis5-7.

In 2019, the American College of Rheumatology/Arthritis Foundation recommended, that in severe, active, chronic AU or in the presence of sight-threatening complications, methotrexate (MTX) and a monoclonal antibody Tumor Necrosis Factor inhibitor (TNFi) should be immediately administered8. Biologic drugs act against specific cytokines or their receptors, in order to reduce tissue damage9. Currently, infliximab, and adalimumab are the main TNF inhibitors available for children10 and are used in the treatment of refractory or chronic childhood uveitis 11,12 . Our study aims to analyze the value and outcome of using biologics at Abou el Reesh, Cairo University Hospital, being a main tertiary referral center in Egypt for children with JIA-U.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed JIA according to rheumatological criteria with ocular affection
* Any type of arthritis (oligoarticular, polyarticular, systemic onset, ocular JIA)
* ANA positive or negative
* Uncontrolled uveitis or frequent relapses

Exclusion Criteria:

* Patients without definitive diagnosis as JIA
* JIA patients on biologics without ocular affection (for systemic control) or with uveitis controlled without the use of biologics
* Patients without adequate duration for follow-up (less than 3 months) or lost follow up data
* Patients without available data prior to the start biologics (to compare control of the uveitis)

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
steroids sparing effect of the drug | 24 months
  reduction in the dosage/frequency of topical and systemic steroids
the severity and complications of the uveitis | 24 months
  degree of clinical improvement by clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Mai Nasser, Principal Investigator — KAsrAlaliny
Locations (1):
- Faculty of medicine, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thorne JE, Woreta F, Kedhar SR, Dunn JP, Jabs DA. Juvenile idiopathic arthritis-associated uveitis: incidence of ocular complications and visual acuity loss. Am J Ophthalmol. 2007 May;143(5):840-846. doi: 10.1016/j.ajo.2007.01.033. Epub 2007 Mar 23. PMID 17362866
- [Background] Qian Y, Acharya NR. Juvenile idiopathic arthritis-associated uveitis. Curr Opin Ophthalmol. 2010 Nov;21(6):468-72. doi: 10.1097/ICU.0b013e32833eab83. PMID 20729734
- [Background] Doycheva D, Deuter C, Stuebiger N, Biester S, Zierhut M. Mycophenolate mofetil in the treatment of uveitis in children. Br J Ophthalmol. 2007 Feb;91(2):180-4. doi: 10.1136/bjo.2006.094698. Epub 2006 Jul 6. PMID 16825275
- [Background] Chang PY, Giuliari GP, Shaikh M, Thakuria P, Makhoul D, Foster CS. Mycophenolate mofetil monotherapy in the management of paediatric uveitis. Eye (Lond). 2011 Apr;25(4):427-35. doi: 10.1038/eye.2011.23. Epub 2011 Mar 18. PMID 21423146
- [Background] Angeles-Han ST, Ringold S, Beukelman T, Lovell D, Cuello CA, Becker ML, Colbert RA, Feldman BM, Holland GN, Ferguson PJ, Gewanter H, Guzman J, Horonjeff J, Nigrovic PA, Ombrello MJ, Passo MH, Stoll ML, Rabinovich CE, Sen HN, Schneider R, Halyabar O, Hays K, Shah AA, Sullivan N, Szymanski AM, Turgunbaev M, Turner A, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Screening, Monitoring, and Treatment of Juvenile Idiopathic Arthritis-Associated Uveitis. Arthritis Rheumatol. 2019 Jun;71(6):864-877. doi: 10.1002/art.40885. Epub 2019 Apr 25. PMID 31021511

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT05540743/Prot_SAP_000.pdf